CLINICAL TRIAL: NCT06582420
Title: Pre-hospital Administration of Fibrinogen Concentrate in Patients With Suspected Trauma-Induced Coagulopathy (PAF-TIC)
Brief Title: Pre-hospital Administration of Fibrinogen in Trauma-Induced Coagulopathy
Acronym: PAF-TIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unidade Local de Saude do Arco Ribeirinho (Other Government)
Collaborators: Unidade Local de Saúde de São José (Unknown); Unidade Local de Saúde da Arrábida (Unknown); Unidade Local de Saúde de Santa Maria (Unknown); Unidade Local de Saúde Almada-Seixal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ULSAR2024
Record Dates: First submitted 2024-08-16; First posted 2024-09-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Trauma Induced Coagulopathy
Keywords: Trauma; Coagulopathy; Trauma Induced Coagulopathy; Fibrinogen; Clot
MeSH Terms: conditions — Wounds and Injuries; Hemostatic Disorders | interventions — Fibrinogen

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to receive either standard trauma care or standard trauma care plus administration of fibrinogen concentrate (FC). The standard of care is determined by national guidelines on trauma, elaborated by the National Institute of Medical Emergency and taught to prehospital physicians and nurses at the time of enrollment in prehospital teams to ensure consistency in the treatment of trauma patients nationwide. The patients assigned to the intervention arm will receive the administration of a fixed dose of 4g fibrinogen, as per previous studies.
  FC will be administered on-scene by prehospital teams as soon as possible, ideally within 60 minutes of injury. Randomization will be performed using sequentially numbered, sealed opaque envelopes. Blood samples will be taken at baseline, upon hospital admission, and at 24h after admission to measure fibrinogen levels and other coagulation parameters. At admission, the PTr and TIC score should be calculated.
Who Masked: Participant, Care Provider
Masking Description: Masking will be applied to participants during all the stay and to care providers until randomly opaque envelopes are opened.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard trauma care (Placebo Comparator): Determined by national guidelines on trauma, elaborated by the National Institute of Medical Emergency and taught to prehospital physicians and nurses at the time of enrollment in prehospital teams to ensure consistency in the treatment of trauma patients nationwide .
  Interventions: Drug: Standard trauma care
- Standard trauma care plus administration of fibrinogen concentrate (FC). (Experimental): The patients assigned to the intervention arm will receive the administration of a fixed dose of 4g fibrinogen, as per previous studies.
  Interventions: Drug: Fibrinogen concentrate

INTERVENTIONS:
Drug: Fibrinogen concentrate — Patients will be randomly assigned to receive either standard trauma care or standard trauma care plus administration of FC. The standard of care is determined by national guidelines on trauma, elaborated by the National Institute of Medical Emergency and taught to prehospital physicians and nurses at the time of enrollment in prehospital teams to ensure consistency in the treatment of trauma patients nationwide. The patients assigned to the intervention arm will receive the administration of a fixed dose of 4g fibrinogen, as per previous studies.
  Arms: Standard trauma care plus administration of fibrinogen concentrate (FC).
Drug: Standard trauma care — Patients will be randomly assigned to receive either standard trauma care or standard trauma care plus administration of FC. The standard of care is determined by national guidelines on trauma, elaborated by the National Institute of Medical Emergency and taught to prehospital physicians and nurses at the time of enrollment in prehospital teams to ensure consistency in the treatment of trauma patients nationwide. The patients assigned to the intervention arm will receive the administration of a fixed dose of 4g fibrinogen, as per previous studies.
  Arms: Standard trauma care

SUMMARY:
A prospective, randomized controlled trial of fibrinogen concentrate (FC) plus standard of care versus standard of care alone in adult trauma patients with major bleeding or presumed major bleeding is developed to evaluate the efficacy and safety of prehospital administration of FC in trauma patients with suspected hypofibrinogenemia and active bleeding or presumed to be bleeding.

The main endpoints are:

1. Plasma fibrinogen levels in the first blood sample drawn at the patient's arrival at the trauma room and/or similar emergency bay dedicated to trauma and reanimation above the critical threshold of 2.0 g/l. As fibrinogen decreases early in trauma, its deficiency predicts massive bleeding and death.
2. Administration feasibility of FC within the prehospital setting.

Patients will be randomly assigned to receive either standard trauma care or standard trauma care plus administration of FC.

DETAILED DESCRIPTION:
Pre-hospital Administration of Fibrinogen Concentrate in Patients with Suspected Trauma-Induced Coagulopathy (PAF-TIC)

Introduction Trauma is a leading cause of morbidity and mortality worldwide, with hemorrhage being one of the primary preventable factors contributing to trauma-related deaths. The management of trauma induced coagulopathy (TIC) is a critical aspect of the resuscitation of severely injured patients. Fibrinogen, a key factor in the coagulation cascade, is often rapidly depleted in cases of severe trauma, leading to compromised clot formation and stability. The use of fibrinogen concentrate (FC) in the pre-hospital setting has emerged as a potential intervention to address this issue and improve patient outcomes.

Recent studies have explored the feasibility, efficacy, and safety of administering FC in both prehospital and emergency departments . A randomized feasibility trial demonstrated that early infusion of FC is attainable and can increase plasma fibrinogen concentration during trauma resuscitation, suggesting that larger trials are justified. Similarly, a prospective, randomized, placebo-controlled trial found that prehospital administration of FC improved blood clot stability and protected against early fibrinogen depletion. These findings are supported by a systematic review, which, despite methodological limitations, indicated that FC administration may reduce the need for blood product transfusion.

In a recently published Australian prehospital study, significant coagulopathy was found to develop in 36% of patients transported to trauma centers and could be found in some patients as early as within 30 minutes of injury. Low fibrinogen was the commonest coagulopathy found among trauma patients and was linked to higher in-hospital mortality rates and an increased need for blood transfusions.

Previous retrospective analyses have provided insights into the effects of FC therapy on fibrinogen levels post-trauma, suggesting that FC does not lead to higher fibrinogen levels beyond the natural acute phase response following tissue injury. Goal-directed coagulation management using thromboelastometry-guided administration of FC has also been associated with favorable survival rates, although the need for prospective, randomized trials has been emphasized.

The ongoing debate regarding the optimal method for fibrinogen replacement in traumatic hemorrhage highlights the importance of further research. While some studies have shown improved survival rates at specific time points following FC administration, the overall impact on hospital mortality remains unclear. The targeted use of FC guided by rotational thromboelastometry has been proposed as a rapid and feasible method to replace fibrinogen, but large multicenter randomized controlled trials are needed to provide conclusive evidence.

Considering these findings, developing a protocol for FC use in the prehospital setting for trauma patients is of paramount importance. Such a protocol would potentially set a standard for FC administration, ensure timely and effective management of TIC, improve the chances of survival and recovery for trauma patients, and optimize the use of blood components and blood-derived products.

Objective To evaluate the efficacy and safety of prehospital administration of FC in trauma patients with suspected hypofibrinogenemia and active bleeding or presumed to be bleeding.

Design A prospective, randomized controlled trial of fibrinogen concentrate plus standard of care versus standard of care alone in adult trauma patients with major bleeding or presumed major bleeding.

Setting Prehospital emergency services from university-affiliated hospitals and regional hospital centers, as well as Helicopter Emergency Medical coordinated by the National Institute of Medical Emergency.

Participants Adult trauma patients with major bleeding and shock, defined by Shock Index, and high likelihood of requiring massive transfusion, defined by mTICCS score.

Stratification Stratification ensures that each treatment group (FC vs. placebo) is balanced in terms of trauma severity. This balance is crucial for minimizing bias and confounding, allowing for a clearer assessment of FC's impact on primary outcomes. During the randomization process, participants should be stratified based on their Injury Severity Score (ISS). ISS is a widely used scoring system to assess trauma severity, with higher scores indicating more severe injuries. Stratification can be achieved by categorizing ISS into predefined ranges (e.g., mild: 1-8, moderate: 9-15, severe: >15).

Interventions Patients will be randomly assigned to receive either standard trauma care or standard trauma care plus administration of FC. The standard of care is determined by national guidelines on trauma, elaborated by the National Institute of Medical Emergency and taught to prehospital physicians and nurses at the time of enrollment in prehospital teams to ensure consistency in the treatment of trauma patients nationwide . The patients assigned to the intervention arm will receive the administration of a fixed dose of 4g fibrinogen, as per previous studies.

Safety Monitoring Adverse events, including thromboembolic events, will be monitored and recorded up to 7 days after hospital admission. A Data Safety Monitoring Board (DSMB) will be established to oversee the trial's safety aspects.

Statistical Analysis Descriptive statistics will be used to summarize patient characteristics. The primary and secondary outcomes will be compared between the FC group and standard of care groups using appropriate statistical tests. Subgroup analyses will be performed based on the severity of the injury, baseline fibrinogen levels at admission, and area of lesions.

Statistical Analysis Plan Sample size calculations: By using an effect size of 0.7, a significance level of 0.1, and a power of 0.8, the required sample size is 26 patients per intervention arm, corresponding to a total sample size of 52 patients

Statistical Methods

* Statistics: Summarize the study population's baseline characteristics (e.g., age, gender, and Injury Severity Score). Means and standard deviations will be reported for continuous variables, while frequencies and percentages will be reported for categorical variables.
* Comparative Analysis: For continuous outcomes, independent t-tests or Mann-Whitney U tests will be used depending on the normality of the data. For categorical outcomes (e.g., incidence of thromboembolic events, mortality rates), chi-square tests or Fisher's exact tests will be used.
* Regression Analysis: Multivariate regression models will be applied to adjust for potential confounders and to identify independent predictors of outcomes.
* Survival Analysis: Kaplan-Meier curves will be constructed for survival data, and differences between groups will be assessed using the log-rank test. Cox proportional hazard models will be used to adjust for covariates.

Handling of Missing Data

Missing data will be handled using the following strategies:

* Complete Case Analysis: Initially, analyses will be conducted on complete cases only.
* Multiple Imputation: If the proportion of missing data is significant, multiple imputation techniques will be used to handle missing values, assuming that the data are missing at random (MAR).
* Sensitivity Analysis: Sensitivity analyses will be performed to assess the robustness of the findings to different methods of handling missing data (e.g., complete case analysis, multiple imputation).

Intention-to-Treat Analysis An intention-to-treat (ITT) analysis will be performed to ensure that all randomized participants are included in the analysis according to the group they were originally assigned, regardless of whether they completed the intervention as per protocol. This approach maintains the benefits of randomization and provides an unbiased estimate of the treatment effect.

Interim Analysis

An interim analysis will be conducted when 50% of the participants have been enrolled and followed up for the primary outcome. The purpose of the interim analysis is to:

* Assess the safety and efficacy of the intervention.
* Make decisions regarding the continuation, modification, or termination of the study based on predefined stopping rules.

A DSMB will oversee the interim analysis and will have the authority to recommend stopping the trial if there is clear evidence of benefit or harm.

Subgroup analyses

Subgroup analyses will be performed to evaluate the consistency of the treatment effect across different patient subgroups. These subgroups may include:

* Severity of injury (stratified by Injury Severity Score).
* Baseline fibrinogen levels (e.g., above or below median level).
* Age groups.
* Gender. These analyses will be pre-specified and interpreted with caution to avoid over- interpretation of findings due to multiple comparisons.

Adjustment for Multiple Comparisons To address the issue of multiple comparisons and control the family-wise error rate, the Bonferroni correction will be applied. If there are comparisons, the significance level for each test will be adjusted to α/k. Alternatively, the False Discovery Rate (FDR) method may be used to control for the proportion of false positives among the significant findings.

The Statistical Analysis Plan for the study will provide a comprehensive framework to ensure rigorous and transparent analysis of the data. The plan includes robust methods for handling missing data, performing intention-to-treat analysis, conducting interim and subgroup analyses, and adjusting for multiple comparisons. This thorough approach will help to ensure the reliability and validity of the study findings, contributing to the evidence base for prehospital administration of fibrinogen concentrate in trauma patients.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients at risk of Trauma Induced Coagulopathy (TIC), with major bleeding or presumed to be bleeding, identified by TIC criteria: mTICCS score > 5 or Shock index > 0.8.

Exclusion Criteria:

* Known adverse reactions to fibrinogen concentrate (FC)
* Isolated trauma such as traumatic head injury only
* Need for cardiopulmonary resuscitation (CPR) on the scene or peri-arrest scenarios
* Deep hypothermia
* Age below 18 years
* Pregnancy
* Prothrombin time ratio superior equal or superior to 1.2 (PTr>1.2) at the hospital admission
* Refusal to participate (if the patients are capable of consenting)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma fibrinogen levels | First 30 minutes on hospital arrival
  Plasma fibrinogen levels in the first blood sample drawn at the patient's arrival at the trauma room and/or similar emergency bay dedicated to trauma and reanimation above the critical threshold of 2.0 g/l. As fibrinogen decreases early in trauma, its deficiency predicts massive bleeding and death.
Administration feasibility | Prehospital setting
  Proportion of Patients Successfully Administered Fibrinogen Concentrate within 60 Minutes Post-Injury.
  This assessment aims to measure the proportion of eligible trauma patients who receive fibrinogen concentrate (FC) within 60 minutes of their injury. Feasibility will be determined by rigorously evaluating the time it takes to administer the treatment, adherence to the protocol, and any operational challenges encountered. Data will be meticulously compiled to calculate the average time it takes to administer the treatment, the rate of successful protocol adherence, and to identify common barriers to timely FC administration.

SECONDARY OUTCOMES:
Mortality | Day 7 and day 28
  Defined as the survival status of the patient regardless of the patient's location (hospital, rehabilitation facility, home).
ICU Length of Stay | Up to 90 days
  The total number of days spent in the Intensive Care Unit (ICU) from the time of admission to the time of transfer out of the ICU.
Multiple Organ Failure | Up to 90 days
  Incidence of multiple organ failure. Data on transfusion requirements and complications will be collected.
Change of fibrinogen levels | Day 1
  Change of serum fibrinogen concentration after administration of FC, by measuring serum fibrinogen levels in the blood sample obtained on scene and the fibrinogen levels in the blood sample obtained in the emergency department.
Change of clot stability upon arrival | First 30 minutes on hospital arrival
  Change in blood clot stability upon arrival at the emergency room, as measured by maximum clot firmness in the FIBTEM assay (FIBTEM MCF) comparing both arms after administration of.
Clot Formation | Up to 90 days
  Clot Formation: Utilize the EXTEM A5 and A10 measured by thromboelastometry as early indicators of clot propagation phase, as they both are both early, sensitive and specific assessments of coagulopathy. Normal Extem A5 ranges from 15 to 25 mm and normal Extem A10 ranges from 22 to 34 mm.
Clot Stability | Up to 90 days
  Clot Stability: Utilize the maximum clot firmness (MCF) measured by thromboelastometry (e.g., ROTEM® FIBTEM assay) as a quantitative indicator of clot stability. The normal range for MCF in the FIBTEM assay typically spans from 9 to 25 mm, indicating the clot's adequate structural integrity under physiological conditions. A clinically significant improvement in clot stability, as evidenced by an increase in MCF, is defined by a post-intervention measurement that exceeds the upper limit of the baseline (pre-intervention) range by at least 20%, ensuring the change is beyond normal variability and likely to impact clinical outcomes.
Incidence of Thromboembolic events | Up to 7 days after hospital admission
  Deep Vein Thrombosis (DVT) is defined by clinical symptoms (limb swelling, pain, and/or redness), plus diagnostic confirmation by ultrasound imaging technique (vein incompressibility or direct thrombus visualization). Thrombosis associated to venous manipulation (such as catheter-related thrombosis) is excluded from this analysis.
  Clinically significant Pulmonary Embolism (PE) is defined by the presence of hypoxic respiratory failure plus the demonstration of a clot in pulmonary arteries by computed tomographic pulmonary angiography (CTPA). Fat or air embolism will be excluded from this analysis.
  Ischemic Stroke diagnosis is defined as the sudden onset of neurological deficits, plus brain ischemia on brain computed tomography (CT) or magnetic resonance imaging (MRI).
  Myocardial Infarction (MI) is defined by chest pain, acute and typical changes on the electrocardiogram (ECG), and elevated cardiac biomarkers like troponin.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Batarda Sena, MD, Principal Investigator — Unidade Local de Saude do Arco Ribeirinho; Francisco Das Neves Coelho, MD, Principal Investigator — Unidade Local de Saude do Arco Ribeirinho; Tiago Quaresma, MD, Principal Investigator — Unidade Local de Saude do Arco Ribeirinho

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Winearls J, Wullschleger M, Wake E, Hurn C, Furyk J, Ryan G, Trout M, Walsham J, Holley A, Cohen J, Shuttleworth M, Dyer W, Keijzers G, Fraser JF, Presneill J, Campbell D. Fibrinogen Early In Severe Trauma studY (FEISTY): study protocol for a randomised controlled trial. Trials. 2017 May 26;18(1):241. doi: 10.1186/s13063-017-1980-x. PMID 28549445
- [Background] Lucena LS, Rodrigues RDR, Carmona MJC, Noronha FJD, Oliveira HP, Lima NM, Pinheiro RB, Silva WAD, Cavalcanti AB. Early administration of fibrinogen concentrate in patients with polytrauma with thromboelastometry suggestive of hypofibrinogenemia: A randomized feasibility trial. Clinics (Sao Paulo). 2021 Nov 8;76:e3168. doi: 10.6061/clinics/2021/e3168. eCollection 2021. PMID 34755760
- [Background] Ziegler B, Bachler M, Haberfellner H, Niederwanger C, Innerhofer P, Hell T, Kaufmann M, Maegele M, Martinowitz U, Nebl C, Oswald E, Schochl H, Schenk B, Thaler M, Treichl B, Voelckel W, Zykova I, Wimmer C, Fries D; FIinTIC study group. Efficacy of prehospital administration of fibrinogen concentrate in trauma patients bleeding or presumed to bleed (FIinTIC): A multicentre, double-blind, placebo-controlled, randomised pilot study. Eur J Anaesthesiol. 2021 Apr 1;38(4):348-357. doi: 10.1097/EJA.0000000000001366. PMID 33109923
- [Background] Aubron C, Reade MC, Fraser JF, Cooper DJ. Efficacy and safety of fibrinogen concentrate in trauma patients--a systematic review. J Crit Care. 2014 Jun;29(3):471.e11-7. doi: 10.1016/j.jcrc.2013.12.011. Epub 2013 Dec 30. PMID 24508201
- [Background] Bodnar D, Bosley E, Raven S, Williams S, Ryan G, Wullschleger M, Lam AK. The nature and timing of coagulation dysfunction in a cohort of trauma patients in the Australian pre-hospital setting. Injury. 2024 Jan;55(1):111124. doi: 10.1016/j.injury.2023.111124. Epub 2023 Oct 14. PMID 37858445
- [Background] Innerhofer N, Treichl B, Rugg C, Fries D, Mittermayr M, Hell T, Oswald E, Innerhofer P, On Behalf Of The Retic Study Group. First-Line Administration of Fibrinogen Concentrate in the Bleeding Trauma Patient: Searching for Effective Dosages and Optimal Post-Treatment Levels Limiting Massive Transfusion-Further Results of the RETIC Study. J Clin Med. 2021 Aug 31;10(17):3930. doi: 10.3390/jcm10173930. PMID 34501379
- [Background] Schochl H, Nienaber U, Hofer G, Voelckel W, Jambor C, Scharbert G, Kozek-Langenecker S, Solomon C. Goal-directed coagulation management of major trauma patients using thromboelastometry (ROTEM)-guided administration of fibrinogen concentrate and prothrombin complex concentrate. Crit Care. 2010;14(2):R55. doi: 10.1186/cc8948. Epub 2010 Apr 7. PMID 20374650
- [Background] Wafaisade A, Lefering R, Maegele M, Brockamp T, Mutschler M, Lendemans S, Banerjee M, Bouillon B, Probst C; Trauma Registry of DGU. Administration of fibrinogen concentrate in exsanguinating trauma patients is associated with improved survival at 6 hours but not at discharge. J Trauma Acute Care Surg. 2013 Feb;74(2):387-3; discussion 393-5. doi: 10.1097/TA.0b013e31827e2410. PMID 23354229
- [Background] Seebold JA, Campbell D, Wake E, Walters K, Ho D, Chan E, Bulmer AC, Wullschleger M, Winearls J. Targeted fibrinogen concentrate use in severe traumatic haemorrhage. Crit Care Resusc. 2019 Sep;21(3):171-178. PMID 31462204
- [Background] Nascimento B, Callum J, Tien H, Peng H, Rizoli S, Karanicolas P, Alam A, Xiong W, Selby R, Garzon AM, Colavecchia C, Howald R, Nathens A, Beckett A. Fibrinogen in the initial resuscitation of severe trauma (FiiRST): a randomized feasibility trial. Br J Anaesth. 2016 Dec;117(6):775-782. doi: 10.1093/bja/aew343. PMID 27956676
- [Background] Kelly JM, Rizoli S, Veigas P, Hollands S, Min A. Using rotational thromboelastometry clot firmness at 5 minutes (ROTEM(R) EXTEM A5) to predict massive transfusion and in-hospital mortality in trauma: a retrospective analysis of 1146 patients. Anaesthesia. 2018 Sep;73(9):1103-1109. doi: 10.1111/anae.14297. Epub 2018 Apr 16. PMID 29658985
- [Background] Blayney A, McCullough J, Wake E, Walters K, Campbell D, Ho D, Chan E, Chalasani A, Winearls J. Substitution of ROTEM FIBTEM A5 for A10 in trauma: an observational study building a case for more rapid analysis of coagulopathy. Eur J Trauma Emerg Surg. 2022 Apr;48(2):1077-1084. doi: 10.1007/s00068-021-01652-w. Epub 2021 Jun 16. PMID 34136958
- [Background] Yurashevich M, Rosser M, Small M, Grotegut C, Kota N, Toffaletti J, Allen T. Evaluating the Association Between Fibrinogen and Rotational Thromboelastometry and the Progression to Severe Obstetric Hemorrhage. Clin Appl Thromb Hemost. 2023 Jan-Dec;29:10760296231175089. doi: 10.1177/10760296231175089. PMID 37186763
- [Background] Hayakawa M. Dynamics of fibrinogen in acute phases of trauma. J Intensive Care. 2017 Jan 20;5(1):3. doi: 10.1186/s40560-016-0199-3. PMID 34798699
- [Background] Okada A, Okada Y, Inoue M, Narumiya H, Nakamoto O. Lactate and fibrinogen as good predictors of massive transfusion in postpartum hemorrhage. Acute Med Surg. 2019 Oct 14;7(1):e453. doi: 10.1002/ams2.453. eCollection 2020 Jan-Dec. PMID 31988765
- [Background] Cho ES, McClelland PH, Cheng O, Kim Y, Hu J, Zenilman ME, D'Ayala M. Utility of d-dimer for diagnosis of deep vein thrombosis in coronavirus disease-19 infection. J Vasc Surg Venous Lymphat Disord. 2021 Jan;9(1):47-53. doi: 10.1016/j.jvsv.2020.07.009. Epub 2020 Jul 30. PMID 32738407
- [Background] Soye JA, Loughrey CB, Hanley PD. Computed tomography pulmonary angiography: a sample of experience at a District General Hospital. Ulster Med J. 2008 Sep;77(3):175-80. PMID 18956799
- [Background] Prisco D, Grifoni E. The role of D-dimer testing in patients with suspected venous thromboembolism. Semin Thromb Hemost. 2009 Feb;35(1):50-9. doi: 10.1055/s-0029-1214148. Epub 2009 Mar 23. PMID 19308893
- [Background] Hasan TF, Hasan H, Kelley RE. Overview of Acute Ischemic Stroke Evaluation and Management. Biomedicines. 2021 Oct 16;9(10):1486. doi: 10.3390/biomedicines9101486. PMID 34680603